CLINICAL TRIAL: NCT01837836
Title: Effect of Health Education on Water Handling Practices in Rural Pondicherry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sri Manakula Vinayagar Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Arun Ghorpade, Assistant Professor, Sri Manakula Vinayagar Medical College and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IEC-49/2012
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Drinking Water Handling Practice; Knowledge of Water Borne Diseases; Bacteriological Quality of Water
Keywords: Health education; water handling practices; Bacteriological quality of water
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Health education (Experimental): The arm includes all the villages under study. Health education will be provided targeting following groups: 1. Home makers 2. School children 3. Water tank operators.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Health education — Health education will include 1. Importance and demonstration of hygienic practices for safe drinking water 2. Promotion of water purification 3. Capacity building of community for safe water availability.

SUMMARY:
The purpose of this study is to assess the drinking water handling practices at household level and to determine the effect of health education on the drinking water handling. Participants from study villages, mainly homemakers, school children and water tank operators who are willing to participate, will be targeted.

Baseline assessment of household practices related to water will be done. Followed by a health education regarding the healthy practices will be given to them. Practice of household water chlorination will be promoted. The healthy behavior will be reinforced through reminders and community activities of self help groups for one year.

The study participants will be benefited from survey in terms of

1. Improved knowledge and practices of drinking water handling
2. Risk reduction of water borne illness to family members

ELIGIBILITY:
Inclusion Criteria:

* Subjects of five study villages

Exclusion Criteria:

* Those who anticipate to move out of study area in next one year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects following hygienic drinking water handling practices | Outcome measure will be assessed at baseline and after one year of health education intervention.

SECONDARY OUTCOMES:
Number of subjects with improved knowledge and practices related to water borne illnesses | Outcome measure will be assessed at baseline and after one year of health education intervention.

OTHER OUTCOMES:
Number of household drinking water samples with improved bacteriological quality | Outcome measure will be assessed at baseline and after one year of health education intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arun G Ghorpade, MD, Principal Investigator — Sri Manakula Vinayagar Medical College and Hospital, Pondicherry
Locations (1):
- Sri Manakula Vinayagar Medical College and Hospital, Puducherry, Puducherry, India